CLINICAL TRIAL: NCT04859868
Title: Non-pharmaceutical Motion Sickness Mitigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gaurav N. Pradhan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20-005763; 80NSSC21K0175 (Other Grant/Funding Number: National Aeronautics and Space Administration)
Record Dates: First submitted 2021-04-01; First posted 2021-04-26 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Subjects attend four visits of the experiment on four separate days. Each visit will be an hour and a half long. In the first visit, subjects will perform batteries of tests that involve balance, cognition, and determine motion perception at different current levels using a rotating chair. In the next three visits, researchers will test the Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair be either turning stimulation ON from beginning, or middle or by not turning ON (the order will be randomized).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Galvanic Vestibular Stimulation During the Entire Session (Experimental): Subjects given Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation ON from beginning.
  Interventions: Device: Galvanic Vestibular Stimulation
- No Galvanic Vestibular Stimulation (No Intervention): Subjects were not given Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation entire session.
- Galvanic Vestibular Stimulation Starting From Mid-session (Experimental): Subjects given Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation ON from the middle of the session.
  Interventions: Device: Galvanic Vestibular Stimulation

INTERVENTIONS:
Device: Galvanic Vestibular Stimulation — Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
  Arms: Galvanic Vestibular Stimulation During the Entire Session; Galvanic Vestibular Stimulation Starting From Mid-session

SUMMARY:
The purpose of this study is evaluate the effect of timing and magnitude on the administration of our nonpharmaceutical treatment to motion sickness, and to evaluate the effect of Galvanic Vestibular Stimulation (GVR) amplitude on functional fitness task performance.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to consent to participate themselves.
* Must be able to attend in-person sessions at the Mayo Aerospace Medicine and Vestibular Research Laboratory in Scottsdale, AZ.
* No racial ethnic groups will be excluded.
* Must be fluent speakers of English.

Exclusion Criteria:

* History of vestibular disease, migraine, or significant balance disorder.
* Traumatic brain injury.
* Recent middle ear infection or recent motion sickness (within 72 hours).
* History of severe motion sensitivity.
* Women who are pregnant.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav N Pradhan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 29 participants were enrolled to receive all interventions, however the order the intervention was received was randomized. All subjects completed the first experimental visit. 2 subjects withdrew from the study prior to the start of the second experimental visit.
Groups:
- GVS Entire Session, GVS From Mid-Session, Then No GVS: Subjects received Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation ON from beginning for experimental visit 1; subjects received GVS ON from mid-session in the rotating chair for experimental visit 2; subjects received GVS stimulation OFF for entire session in rotating chair for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
- GVS Entire Session, No GVS, Then GVS From Mid-Session: Subjects received Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation ON from beginning for experimental visit 1; subjects received GVS stimulation OFF for entire session in rotating chair for experimental visit 2; subjects received GVS ON from mid-session in the rotating chair for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
- GVS From Mid-Session, GVS Entire Session, Then No GVS: Subjects received Galvanic Vestibular Stimulation (GVS) ON from mid-session in the rotating chair for experimental visit 1; subjects received GVS to mitigate motion sickness in the rotating chair turning stimulation ON from beginning for experimental visit 2; subjects received GVS stimulation OFF for entire session in rotating chair for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
- GVS From Mid-Session, No GVS, Then GVS Entire Session: Subjects received Galvanic Vestibular Stimulation (GVS) ON from mid-session in the rotating chair for experimental visit 1; subjects received GVS stimulation OFF for entire session in rotating chair for experimental visit 2; subjects received GVS to mitigate motion sickness in the rotating chair turning stimulation ON from beginning for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
- No GVS, GVS From Mid-Session, Then GVS Entire Session: Subjects received Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation OFF from beginning for experimental visit 1; subjects received GVS ON from mid-session in the rotating chair for experimental visit 2; subjects received GVS stimulation ON for entire session in rotating chair for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
- No GVS, GVS Entire Session, Then GVS From Mid-Session: Subjects received Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair turning stimulation OFF from beginning for experimental visit 1; subjects received GVS stimulation ON for entire session in rotating chair for experimental visit 2; subjects received GVS ON from mid-session in the rotating chair for experimental visit 3.
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
Period: First Experimental Visit (1.5 Hour)
Arm/Group | GVS Entire Session, GVS From Mid-Session, Then No GVS | GVS Entire Session, No GVS, Then GVS From Mid-Session | GVS From Mid-Session, GVS Entire Session, Then No GVS | GVS From Mid-Session, No GVS, Then GVS Entire Session | No GVS, GVS From Mid-Session, Then GVS Entire Session | No GVS, GVS Entire Session, Then GVS From Mid-Session
Started | 5 | 5 | 5 | 4 | 5 | 5
Completed | 5 | 5 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Experimental Visit (1.5 Hour)
Arm/Group | GVS Entire Session, GVS From Mid-Session, Then No GVS | GVS Entire Session, No GVS, Then GVS From Mid-Session | GVS From Mid-Session, GVS Entire Session, Then No GVS | GVS From Mid-Session, No GVS, Then GVS Entire Session | No GVS, GVS From Mid-Session, Then GVS Entire Session | No GVS, GVS Entire Session, Then GVS From Mid-Session
Started | 4 | 5 | 5 | 4 | 4 | 5
Completed | 4 | 5 | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Experimental Visit (1.5 Hour)
Arm/Group | GVS Entire Session, GVS From Mid-Session, Then No GVS | GVS Entire Session, No GVS, Then GVS From Mid-Session | GVS From Mid-Session, GVS Entire Session, Then No GVS | GVS From Mid-Session, No GVS, Then GVS Entire Session | No GVS, GVS From Mid-Session, Then GVS Entire Session | No GVS, GVS Entire Session, Then GVS From Mid-Session
Started | 4 | 5 | 5 | 4 | 4 | 5
Completed | 4 | 5 | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Galvanic Vestibular Stimulation: Subjects attend four visits of the experiment on four separate days. Each visit will be an hour and a half long. In the first visit, subjects will perform batteries of tests that involve balance, cognition, and determine motion perception at different current levels using a rotating chair. In the next three visits, researchers will test the Galvanic Vestibular Stimulation (GVS) to mitigate motion sickness in the rotating chair be either turning stimulation ON from beginning, or middle or by not turning ON (the order will be randomized).
  Galvanic Vestibular Stimulation: Low electrical currents to the vestibular system, to induce the realistic sensation of motion (i.e., the g-forces that occur during flight) as well as null out motion perception.
Arm/Group | Galvanic Vestibular Stimulation
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Motion Perception
Description: Motion Perception verbal report using a visual analog scale (1-100) will be recorded during the rotation of the chair (1=feeling no motion perception; 100=feeling the maximum motion perception)
Time Frame: During the rotation of the chair, approximately 1 hr
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galvanic Vestibular Stimulation
Number analyzed (Participants) | 27
score on a scale
  No GVS | 55.3 (32.2)
  GVS Entire Session | 49.7 (34.0)
  GVS from Mid-Session | 50.1 (33.6)

2. Secondary Outcome: Motion Sickness Questionnaire
Description: subjective experiences of motion sickness in a scale of 0-10 (0=not at all; 10=most severe)
Time Frame: During the rotation of the chair, approximately 1 hr
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galvanic Vestibular Stimulation
Number analyzed (Participants) | 27
score on a scale
  No GVS | 3.0 (2.9)
  GVS Entire Session | 3.2 (3.2)
  GVS from Mid-Session | 3.4 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 4 days on all participants.
Arm/Group | Galvanic Vestibular Stimulation During the Entire Session | No Galvanic Vestibular Stimulation | Galvanic Vestibular Stimulation Starting From Mid-session
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT04859868/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04859868/ICF_001.pdf